CLINICAL TRIAL: NCT07172659
Title: A 12-week, Open-label, Randomized, Standard of Care Controlled, Dose-ranging Safety and Efficacy Study of Dovramilast in People With Moderate to Severe Acute or Recurrent Leprosy Type 2 Reaction
Brief Title: Efficacy and Safety Study of Dovramilast in People With Leprosy Type 2 Reaction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDGH-DOV-2001
Record Dates: First submitted 2025-08-07; First posted 2025-09-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Erythema Nodosum Leprosum
Keywords: Leprosy type 2 reaction; dovramilast
MeSH Terms: interventions — Prednisolone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dovramilast 100 mg (Experimental)
  Interventions: Drug: Dovramilast
- Dovramilast 150 mg (Experimental)
  Interventions: Drug: Dovramilast
- Standard of care (Active Comparator): Prednisolone (or thalidomide US sites only)
  Interventions: Drug: Prednisolone; Drug: Thalidomide

INTERVENTIONS:
Drug: Dovramilast — Dovramilast
  Arms: Dovramilast 100 mg; Dovramilast 150 mg
Drug: Prednisolone — Standard of care
  Arms: Standard of care
Drug: Thalidomide — Standard of care (US only)
  Arms: Standard of care

SUMMARY:
Dovramilast has not been approved for leprosy type 2 reaction (erythema nodosum leprosum, ENL) or any other disease anywhere in the world. In this study, an experimental drug called dovramilast is being tested to see how it compares to current treatments for leprosy type 2 reaction. Specifically, this study aims to assess the efficacy of 100mg or 150 mg dovramilast compared with standard treatments (also known as standard of care). This study also aims to assess the safety of two strengths in adults with leprosy type 2 reaction.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years of age or older.
2. Provision of written informed consent.
3. Laboratory confirmed previous or current Mycobacterium leprae or Mycobacterium lepromatosis infection.
4. Leprosy type 2 reaction meeting the following criteria:

   * Either:

     i. Acute (first episode and no treatment initiated) or ii. Recurrent (at least one further episode occurring 28 days or more after withdrawal of leprosy type 2 reaction treatment).
   * Presence of at least 10 leprosy type 2 reaction tender papular and/or nodular skin lesions (not including scars).
   * An ENLIST score of at least 9.
5. If a woman of reproductive potential, agree to the use of two reliable contraceptive measures (at least one of which is a highly effective form of contraception) from Screening until at least 4 weeks after completion of treatment with dovramilast or standard of care. Refer to Special Considerations for additional information.
6. If male (including those who have had a successful vasectomy), agree to using a latex condom during any sexual contact with women of reproductive potential from Screening until at least 4 weeks after completion of treatment with dovramilast or standard of care.

Exclusion Criteria:

1. Chronic leprosy type 2 reaction, defined as the reaction occurring for 24 weeks or more during which a subject has required treatment either continuously or where any treatment free period had been < 28 days.
2. Receipt of thalidomide, lenalidomide, pomalidomide, systemic corticosteroids, clofazimine (> 50 mg/day), apremilast or any other phosphodiesterase (PDE) 4 inhibitor, or immunosuppressive/immunomodulatory treatment within 28 days of Baseline.
3. Receipt of an investigational agent within 28 days of Baseline or 5 half-lives of the investigational agent (whichever is longer).
4. Leprosy type 2 reaction with orchitis, uveitis, iritis, or severe neuritis (Grade 3 or greater severe neuritis).
5. Current diagnosis of leprosy type 1 reaction or Lucio's phenomenon.
6. Current tuberculosis, malaria, cutaneous or visceral leishmaniasis or other serious bacterial, viral, or parasitic infection at Screening or Baseline.
7. Active systemic fungal infection requiring or undergoing treatment.
8. Other than leprosy type 2 reaction, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
9. Other than leprosy type 2 reaction, any other dermatological condition that could, in the opinion of the Investigator, interfere with the study assessments.
10. Chronic hepatitis B, chronic hepatitis C, or human immunodeficiency virus (HIV) positive.
11. Pregnant women or breastfeeding mothers.
12. Use (or planned use) of antimetabolites or alkylating agents, rifampin use more frequent than monthly, phenobarbital, carbamazepine, phenytoin, traditional or herbal preparations (including St. John's wort), foods (including grapefruit) known to affect activity of the cytochrome (CYP)3A4 enzyme or use (or planned use) of all strong CYP3A and P-gp inhibitors including ketoconazole, itraconazole, voriconazole, posaconazole, clarithromycin, ritonavir, cobicistat, diltiazem. Substrates of CYP3A4, CYP2C9, CYP2C19, and P-gp should be used with caution when concomitantly administered with dovramilast.
13. Known or suspected active substance abuse or a history of substance abuse within 6 months prior to Screening.
14. Prior history of suicide attempt at any time in the subject's lifetime prior to Screening or Randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
15. Current diagnosis of depression, and/or history of suicide ideation
16. History of or presence of cardiac disease, including:

    * Clinically significant abnormal electrocardiogram
    * QTcF > 450 msec
17. Receipt of a vaccination within 7 days of Baseline.
18. Known or suspected hypersensitivity to: PDE4 inhibitors including dovramilast or apremilast; thalidomide; prednisolone, or; excipients used in the formulation of dovramilast, thalidomide or prednisolone.
19. Body Mass Index < 15 kg/m^2 or > 35 kg/m^2.
20. Unable to, or significant difficulty with, swallowing tablets/capsules.
21. Anemia requiring transfusion.
22. History of or current pancreatitis.
23. Known or suspected cirrhosis of the liver.
24. The following laboratory abnormalities:

    * White blood cells (WBC) < 2.5 x 10^9/ L.
    * Neutrophils (granulocytes) < 1.0 x 10^9/L.
    * Platelets < 80 x 10^9/L.
    * Aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of reference range.
    * Albumin < 30 mg/dL.
    * Bilirubin > 2 mg/dL
    * Calculated creatinine clearance (Cockcroft Gault) < 50 milliliter (mL)/minute.
    * Lipase ≥ 1.6 times the upper limit
25. Previous participation in this study
26. Unwilling, unlikely or unable to comply with all protocol specified assessments, including photographic assessments
27. Enrolled in another leprosy type 2 reaction treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of dovramilast (100 mg or 150 mg) recipients achieving a 75% improvement in leprosy type 2 reaction skin lesions at week 12 | 12 weeks
  The proportion of subjects achieving a reduction of leprosy type 2 reaction skin lesion count of at least 75% from Baseline at Week 12 without the need for rescue.
  Rescue is defined as:
  1. A change from dovramilast at any dose to standard of care or dose maintenance beyond taper time points defined in standard of care treatment guidelines (and specified in this protocol), or
  2. Standard of care dose increase, switching to or adding another leprosy type 2 reaction treatment
Incidence and severity of adverse events | 12 weeks
  The incidence and severity of adverse events, changes in vital signs and blood dyscrasias

SECONDARY OUTCOMES:
Resolution of fever to ≤ Grade 1 | 12 weeks
  Proportion of subjects with resolution of fever to ≤ Grade 1 among the subgroup of subjects with fever present at Baseline at Grade 2 or greater.
Skin lesion count changes | 12 weeks
  • Change from Baseline in skin lesion count up to and including Week 12.
Change from Baseline ENLIST (Erythema Nodosum Leprosum International Study ) severity scale score | At each post Baseline time point
Change from Baseline of each of the following parameters when present at Baseline at Grade 2 or greater | from baseline to Week 12
  * Leprosy type 2 reaction lesions with respect to: number, inflammation, and extent
  * Neuritis
  * Pain:
  * Fever
  * Peripheral edema with respect to location and severity
  * Inflammation of joints and/or digits
  * Lymphadenopathy
Changes in neuropathy from Baseline grade | 12 weeks
Time to resolution | 12 weeks
  For each individual leprosy type 2 reaction when present at least Grade 1 at Baseline
Proportion of subjects requiring Rescue medication and time to initiation of Rescue medication | 12 weeks
Total amount of treatment for leprosy type 2 reaction administered | 12 weeks
Recurrences | 48 weeks
  Recurrence is defined as new signs and symptoms consistent with leprosy type 2 reaction. The number of Recurrence episodes requiring treatment.
Exposure metrics of dovramilast | 48 weeks
  Area under the curve (AUC)
Exposure metrics of the dovramilast metabolite M15 | 48 weeks
  Area under the curve (AUC)
Skin lesion count changes | 12 weeks
  • Proportion of Responders at each post-Baseline timepoint.
Skin lesion count changes | 12 weeks
  Proportion of subjects achieving a reduction of leprosy type 2 reaction skin lesion count from Baseline of 50%, 90% and 100% without Rescue at Week 12.
Exposure metrics of dovramilast | 48 weeks
  Including AUC, Cmax, and Tmax.
Exposure metrics of dovramilast | 48 weeks
  Cmax
Exposure metrics of dovramilast | 48 weeks
  Tmax.

OTHER OUTCOMES:
Quantification of immunological markers in whole blood samples by central laboratory, blinded to patient identification, treatment arm, and study visit | 48 weeks
  Concentration of inflammatory cytokines
Quantification of immunological markers in skin biopsies by central laboratory, blinded to patient identification, treatment arm, and study visit | 48 weeks
  Leukocyte infiltration of skin lesions by histology

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Harborview Medical Center, University of Washington, Seattle, Washington
- Centre de Dépistage de Traitement de la Lèpre et de l'Ulcère de Burulli, Abomey-Calavi, Benin
- Chr de Divo, Divo, Côte d’Ivoire
- Universitas Gadjah Mada, Yogyakarta, Indonesia
- Philippine General Hospital, University of the Philippines, Manila, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Undecided